CLINICAL TRIAL: NCT00645749
Title: Helminth-induced Immunomodulation Therapy (HINT) in Relapsing-remitting Multiple Sclerosis
Acronym: HINT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0484, 2007-0390
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Therapy with Helminths

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Helminth ova (Experimental): Subjects serving as their own controls (baseline - end-of-treatment) will receive a dose of 2,500 ova, in liquid form, every 2 weeks
  Interventions: Biological: Helminth ova

INTERVENTIONS:
Biological: Helminth ova — 2500 ova per dose (liquid form)
  Other Names: Therapy with Helminths

SUMMARY:
The hypothesis of this study is that helminth-induced immunomodulation therapy (HINT) will be safe and effective when administered orally in patients with relapsing-remitting multiple sclerosis (RRMS).

DETAILED DESCRIPTION:
Phase 1 of the HINT trial was completed with enrollment of 5 subjects. HINT Phase 2 is now closed to enrollment of 15 subjects. Recruitment sites are the UW-Madison and the Marshfield Clinic.

ELIGIBILITY:
Inclusion Criteria:

* McDonald Committee (2010) criteria for RRMS (MS) .
* ambulatory patients with disability scores of EDSS 0.-5.0
* male or female subjects; ages 18-50
* diagnosis within three years of study entry, based on either a) two or more clinical attacks in the three years prior to entry or b) one attack within three years of entry, coupled with MRI evidence of dissemination in space and time by strict application of McDonald Committee MRI criteria
* active MRI at entry, as evidenced by at least one gd+ enhancing lesion during screening
* explicit refusal to be treated with conventional disease-modifying medications (DMT) for RRMS, after full discussion of the potential benefits and risks of these agents and after review of the National Multiple Sclerosis Advisory Statement DMT.
* ability to provide written informed consent

Exclusion Criteria:

* patients who are unwilling or unable to give written informed consent or to follow the protocol successfully
* allergy to Trichuris species
* treatment with metronidazole (Flagyl) or other medications with anti-helminth effects (IB 5.7)
* previous or anticipated treatment with FDA-approved or other experimental medications for RRMS
* previous treatment with immunosuppressive therapy, cytotoxic chemotherapy, or lymphoid irradiation for any reason
* insulin dependent diabetes mellitus
* history of HIV-1, HTLV-1, viral hepatitis, or Lyme disease.
* requirement for chronic, sustained aspirin or non-steroidal anti-inflammatory medications (e.g., use of more than 5-6 days per month for transient symptoms)
* significant physical or mental disease which would preclude successful compliance and participation in the study or, in the opinion of the principal investigator, constitute a hazard, such that enrollment in the study would not be in the patient's best interest.
* presence or history of cancer of any type (except successfully treated basal cell or squamous cell carcinoma of skin)
* history of alcohol or drug abuse in last 12 months; chronic liver or biliary disease; AST or ALT determination greater than two times the upper limit of normal
* any of the following laboratory abnormalities: serum creatinine > 1.7 mg/DL, white blood count < 3,500/mm3, lymphocyte count < 800/mm3
* special subjects such as minor children, mentally disabled persons, or prisoners
* any contraindication to MRI scanning, including significant claustrophobia or sensitivity to gadolinium contrast agent
* pregnancy and lactation; women of childbearing potential must have a documented negative serum beta HCG pregnancy test at entry and during the study and must be willing to practice adequate birth control for the duration of the study
* any MS attack or treatment with corticosteroid medication within 30 days of study entry (corticosteroids may be used during the study for MS relapses per the judgment of the treating physician, IB 5.7, IB 6.1.3)
* immediate household or family contacts who are immunodeficient or immunosuppressed
* history of parasitism or positive determination ova and parasite stool at screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-07; Primary Completion 2015-08-13 (Actual); Study Completion 2015-08-13 (Actual)

PRIMARY OUTCOMES:
MS activity, as judged by the number of new gadolinium-enhancing lesions on serial MRI scans | Up to 19 months
  MS activity will be assessed based on the number of new gadolinium-enhancing lesions on serial MRI scans.

CONTACTS AND LOCATIONS:
Overall Officials: John O Fleming, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Fleming J, Hernandez G, Hartman L, Maksimovic J, Nace S, Lawler B, Risa T, Cook T, Agni R, Reichelderfer M, Luzzio C, Rolak L, Field A, Fabry Z. Safety and efficacy of helminth treatment in relapsing-remitting multiple sclerosis: Results of the HINT 2 clinical trial. Mult Scler. 2019 Jan;25(1):81-91. doi: 10.1177/1352458517736377. Epub 2017 Oct 24. PMID 29064315
- [Derived] Fleming JO, Isaak A, Lee JE, Luzzio CC, Carrithers MD, Cook TD, Field AS, Boland J, Fabry Z. Probiotic helminth administration in relapsing-remitting multiple sclerosis: a phase 1 study. Mult Scler. 2011 Jun;17(6):743-54. doi: 10.1177/1352458511398054. Epub 2011 Mar 3. PMID 21372112